CLINICAL TRIAL: NCT01001455
Title: Clinical Test for Armed-used Blood Pressure Monitor With Preformed Cuff
Status: Completed | Type: Observational
Sponsor: Andon Health Co., Ltd (Industry)
Responsible Party: Liu Yi, Andon Health co., LTD
Other Study IDs: AndonHealth3
Record Dates: First submitted 2009-10-23; First posted 2009-10-26 (Estimated); Last update posted 2009-10-26 (Estimated); Status verified 2009-10

CONDITIONS: Blood Pressure
Keywords: BP

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- blood pressure monitor: Cuff circumference:22cm-36cm
- stethoscopy: Cuff circumference: 22cm-36cm

SUMMARY:
The purpose of this study is to monitor the blood pressure level of the patient using a preformed cuff ranged 22 cm-36 cm.

ELIGIBILITY:
Inclusion Criteria:

* cuff circumference:22cm-36cm

Exclusion Criteria:

* None

Ages: 23 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: resident of a community.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2009-08; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
level of blood pressure | 10S